CLINICAL TRIAL: NCT06220500
Title: Radiomics Analysis Based on MRI to Detect Brucella Spondylitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Inner Mongolia Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: AHInnerMongolia-BS
Record Dates: First submitted 2024-01-11; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Brucella Spondylitis
Keywords: Radiomics; MRI

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Brucella spondylitis, an infectious spinal disease caused by the invasion of Brucella bacteria into the body. Its diagnosis relies mainly on laboratory and imaging tests. Due to the limited diagnostic ability of X-ray and CT for Brucella spondylitis, MRI has become the main diagnostic tool. In recent years, functional magnetic resonance technology has demonstrated great advantages in the diagnosis and therapeutic evaluation of brucellosis spondylitis, which can provide pathophysiologic information about the disease and is also a noninvasive and noninvasive diagnostic tool with a broader application prospect. Radiomics, an emerging approach, has also shown better diagnostic efficacy for this disease.

DETAILED DESCRIPTION:
The investigators will incorporate 100 confirmed cases of Brucella spondylitis (BS) patients diagnosed at Affiliated Hospital of Inner Mongolia Medical University. The patients receive routine scan with a Siemens Skyra 3.0T MRI scanner and the investigators collect clinical data and blood test results from the patients.The investigators segment the affected vertebral bodies by ITK-SNAP software on STIR images to create three-dimensional regions of interest. Then use Onekey software to extract radiomics features from the affected vertebral bodies. Employed t-tests and Lasso regression to select radiomics features. Then separately use radiomics features and combining it with clinical information to build random vector machine(SVM) and random forest(RF) models . All the models are constructed in the training set and their performance are evaluated on the validation set.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients/Inpatients
2. Age 18-70 years
3. Meet diagnostic criteria for brucellosis
4. Meet symptoms of brucellosis spondylitis
5. Voluntarily sign an informed consent form
6. Can cooperate with MRI examination

Exclusion Criteria:

1. Patients with serious diseases of other systems
2. History of malignant tumors of the vertebral body
3. History of tuberculosis
4. Contraindications to magnetic resonance imaging

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: About 100 patients with Brucellosis including patients with brucella spondylitis obviously and patients with obvious waist pain and the conventional MRI showed abnormalities were selected.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The useful value of radiomics of MRI in BS clinical diagnosis. | December 2024
  The investigators will validate the results. The validation and external test cohorts will be used to evaluate the performance of the prediction models. The micro-avg and macro-avg precision, true positive (TP), true negative (TN), false positive (FP), false negative (FN), accuracy, sensitivity, specificity, and F1 score of different models will be calculated. Receiver operating characteristic (ROC) curves is going to be used to assess the sensitivity and specificity of the models, and the area under the ROC curve (AUC) was used to describe the discriminative power of the models. The investigators think radiomics of MRI can provide a reliable basis for early damage in brucellosis spondylitis and provides evidence for early clinical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Peng fei Qiao, MD, Study Director — The Affiliated Hospital of Inner Mongolia Medical University
Locations (1):
- Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia, China